CLINICAL TRIAL: NCT04010643
Title: Clinical and Economic Evaluation of Neurocognitively-Enhanced Online Cognitive Behavioural Therapy to Promote Functional Recovery Among Community-Living Individuals With Depression: OPTM Study (Online Psychological Treatments for Low Mood)
Brief Title: Clinical and Economic Evaluation of Neurocognitively-Enhanced Online Cognitive Behavioural Therapy
Acronym: OPTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Irish Research Council (Other); Inštitut za ekonomska raziskovanja (Institute for Economic Research, Slovenia) (Unknown); University of Limerick (Other)
Responsible Party: Principal Investigator, Maria Semkovska, Principal Investigator of OPTM Study, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDU_MS_02
Record Dates: First submitted 2019-06-22; First posted 2019-07-08 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Depression
Keywords: online cognitive behavioural therapy; online neurocognitive remediation; memory; sustained attention; everyday occupational function; economic evaluation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The study will be a two-group parallel-design randomised controlled trial comparing online cognitive behavioural therapy (oCBT) to oCBT enhanced with neurocognitive remediation for depression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online cognitive behavioural therapy (oCBT) (Active Comparator): 20 hours of online engagement with the oCBT programme over 5 weeks, distributed as follows.
  Each week, the participants complete 1 hour of of the MoodGym program, followed by 2 hours of practical online CBT homework. To equate time and type of engagement spent in doing oCBT and oCBT+NCRT, 1 final hour per week is dedicated to completing online puzzles.
  Interventions: Behavioral: online cognitive behavioural therapy
- online neurocognitively-enhanced CBT (oCBT+oNCRT) (Experimental): 20 hours of online engagement with the oCBT+oNCRT programme over 5 weeks, distributed as follows.
  Each week, the participants complete 1 hour of the MoodGym program, followed by 1 hour of practical online CBT homework & 3 hours of the online NCRT programme Cognifit targeting attention, memory, and planning ability.
  Interventions: Behavioral: online cognitive behavioural therapy; Behavioral: online neurocognitive remediation therapy

INTERVENTIONS:
Behavioral: online cognitive behavioural therapy — oCBT: MoodGym is a 5-week oCBT program developed by the Centre for Mental Health Research at the Australian National University. This program has been shown to be clinically effective at reducing mood symptoms in depression studies (see meta-analytical review of Twomey & O'Reilly, 2017). MoodGym consists of a number of interactive modules to be completed sequentially and including work on own feelings, thoughts, methods to change dysfunctional thinking patterns, de-stressing, and relaxation. Each module is followed by an associated practical homework, while a personalised workbook allows the participant to track their mood profile and progress throughout the modules.
Behavioral: online neurocognitive remediation therapy — NCRT involves the behavioural application of structured exercises targeting neurocognitive processes by mobilising neuroplasticity that is the brain's ability to adjust its function in response to environmental change. Computerised NCRT has demonstrated efficacy to improve attention, working memory and global functioning in depression (Motter et al., 2016; Semkovska et al., 2015). NCRT is delivered through the Cognifit online programme. The Cognifit modules were selected as targeting remediation of neurocognitive domains known to be impaired in depression, i.e. selective and divided attention, visual and verbal working memory, and everyday planning (Hammar and Ardal, 2009; Semkovska et al., 2019).
  Arms: online neurocognitively-enhanced CBT (oCBT+oNCRT)

SUMMARY:
To evaluate the clinical efficacy of online cognitive behavioural therapy supplemented with online neurocognitive remediation therapy to improve mood and cognition, decrease relapse rates and optimise work and occupational functioning.

DETAILED DESCRIPTION:
Depression is the most prevalent mental disorder with high relapse rates. Direct costs to Europe represent 1% of its total economy. Following usual treatment, mood improves or fully recovers but cognitive deficits often persist, preventing full return to normal social function. These deficits worsen with repeated depressive episodes and are a significant predictor of relapse. Preventing depression relapse remains one of the biggest therapeutic challenges in the field. While effective short-term therapies, such as cognitive behavioural therapy (CBT), exist, all are associated with high relapse rates. Online neurocognitive remediation therapy (oNCRT), by its potential to rehabilitate impaired cognition in depression, offers an innovative solution to this mental health problem.

This trial aims to test the effectiveness and cost-effectiveness of neurocognitively enhanced online CBT to improve mood and cognition in depression, optimise everyday functioning and prevent depression relapse over six months follow-up, using a randomised active-control parallel-groups research design. Individuals presenting with at least mild depression (n=134) are randomly assigned to one of two treatment allocations: online CBT (oCBT) or neurocognitively enhanced online CBT (oCBT+oNCRT) for 20 one-hour sessions over 5 weeks (i.e., four weekly sessions).

Before randomisation and within a week of the final allocated session, mood, attention, memory and planning abilities will be assessed. All participants will be then followed for six-months to determine if the mood and cognitive benefits of the oCBT+oNCRT are maintained with the passage of time compared to the control group (oCBT alone). Standard measures of daily functioning (e.g., work ability, occupational function) and economic cost-effectiveness data will be obtained at the same time points. Demonstrating the oNCRT effectiveness as an adjunct to CBT will contribute towards optimising connected healthcare solutions for depression.

ELIGIBILITY:
Inclusion Criteria:

* scoring a minimum of 14 on the BDI-II,
* internet access
* computer access
* English-speaking fluency

Exclusion Criteria:

* scoring less than 14 on BDI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms at end of treatment | through study completion, an average of 1 year
  The Beck's Inventory for Depression - II (BDI-II; Beck et al., 1996) assesses the self-report severity of currently experienced depressive symptoms. The total score of 21 items is used.The scale score ranges 0 to 63, with higher values indicating more severe depression. Scores are to be interpreted as follows: 0-8: no depression; 9-13: subsyndromal depressive symptoms; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Relapse rates at 6 months follow-up | through study completion, an average of 1 year
  Percent individuals, whose Beck's Inventory for Depression - II score at end of treatment was below 14, but returned to above 14 at 6-months follow-up

SECONDARY OUTCOMES:
Immediate verbal memory (cognitive outcome 1) | through study completion, an average of 1 year
  will be assessed with the Logical Memory, a standardized neuropsychological test assessing the ability to recall two stories that one has just heard (Lezak et al., 2012) and after a delay. The first part (Logical memory I) measures immediate verbal memory, with total score ranging 0 to 75, with higher values suggesting better memory
Delayed verbal memory (cognitive outcome 2) | through study completion, an average of 1 year
  will be assessed with the Logical Memory, a standardized neuropsychological test assessing the ability to recall two stories that one has just heard (Lezak et al., 2012) and after a delay. The first part (Logical memory II) measures delayed verbal memory, with total score ranging 0 to 50, with higher values suggesting better memory
Inhibition ability (cognitive outcome 3) | through study completion, an average of 1 year
  will be assessed with the Colour Word Interference Test, a standardized neuropsychological test which third part is designed to assess the individual's ability to inhibit a predominant response (reading a meaningful word) and provide a required response (naming the ink in which a word is printed). Speed of performance (in seconds) at the third part of the test is used to determine inhibition ability, with longer time taken to complete task meaning lower performance.
Flexibility ability (cognitive outcome 4) | through study completion, an average of 1 year
  will be assessed with the Colour Word Interference Test, a standardized neuropsychological test which forth part is designed to assess the individual's ability to flexibly shift between a predominant response (reading a meaningful word) and a non dominant required response (naming the ink in which a word is printed). Speed of performance (in seconds) at the forth part of the test is used to determine flexibility ability, with longer time taken to complete task meaning lower performance.
Verbal working memory (cognitive outcome 5) | through study completion, an average of 1 year
  The Digit Span Backwards neuropsychological test is used to assess verbal working memory. It requires the individual to repeat in reverse order a sequence of numbers. The length of the sequence increases after every second trial. The score range is 0 to 16, with higher scores meaning better verbal working memory
Planning ability (cognitive outcome 6) | through study completion, an average of 1 year
  The Towers neuropsychological test is used to assess planning ability. It requires solving problems of increasing difficulty that involve the reproduction of tower models given a specific set of rules. The score range is 0 to 22, with higher scores meaning better planning ability.
Work and Social Adjustment (occupational outcome 1) | through study completion, an average of 1 year
  will be measured with the Work and Social Adjustment Scale, a 5-item self-report questionnaire assessing the impact of depression on current everyday occupational functioning (Mundt et al., 2002). The score range is 0 to 40, with higher scores meaning lower quality of occupational functioning.
Costs Associated with Mental Healthcare (economic main assessment) | through study completion, an average of 1 year
  Costs Associated with Mental Healthcare Questionnaire, A questionnaire designed to collect data regarding the costs of depression across areas including medication, hospitalisations,consultations with mental healthcare specialists, travel, time away from work etc.; higher values of all items indicate higher costs

OTHER OUTCOMES:
Work Productivity and the Activity (occupational outcome 2) | through study completion, an average of 1 year
  will be measured with the Work Productivity and Activity Impairment Scale, a 6-item self-report questionnaire (Reilly et al., 1993). Each item, with ranges 0 to 10 will be analysed separately, with higher values representing lower work productivity
Health-Related Quality of Life (Economic outcome 2): EQ-5D-5L | through study completion, an average of 1 year
  will be measured with the EQ-5D-5L self-report questionnaire regarding areas of mobility, self-care, usual activities, pain/discomfort, anxiety. Responses allow for the calculation of quality adjusted life years that are used to inform economic evaluations of healthcare (EuroQol Group, 1990), with scores varying from 0 to 25, with higher values meaning lower quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Maria Semkovska, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No